CLINICAL TRIAL: NCT01857206
Title: A Phase III, Observer Blind, Randomized, Controlled, Multicenter Study to Evaluate the Safety of a Trivalent Subunit Influenza Vaccine Produced Either in Mammalian Cell Culture or in Embryonated Chicken Eggs (Fluvirin®), in Healthy Children and Adolescents 4 to 17 Years of Age.
Brief Title: Safety of Two Trivalent Influenza Vaccines Evaluated in Children and Adolescents 4 to 17 Years of Age
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Vaccines (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: V58_31; U1111-1139-9440 (Other: Universal Trial Number (UTN))
Record Dates: First submitted 2013-05-16; First posted 2013-05-20 (Estimated); Results first posted 2014-11-03 (Estimated); Last update posted 2014-12-05 (Estimated); Status verified 2014-11

CONDITIONS: Influenza; Fever
Keywords: Influenza; children and adolescents; trivalent vaccine; cell culture; embryonated chicken eggs
MeSH Terms: conditions — Influenza, Human; Fever

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- TIVc (Experimental): Subjects ≥4 to ≤17 years of age received one or two doses of mammalian cell-culture-derived trivalent influenza vaccine based on their previous vaccination status.
  Interventions: Biological: Mammalian cell based flu vaccine
- TIVf (Active Comparator): Subjects ≥4 to ≤17 years of age received one or two doses of egg-derived trivalent influenza vaccine based on their previous vaccination status.
  Interventions: Biological: Egg based flu vaccine

INTERVENTIONS:
Biological: Mammalian cell based flu vaccine
  Arms: TIVc
Biological: Egg based flu vaccine
  Arms: TIVf

SUMMARY:
Evaluate safety and tolerability of TIVa or TIVb vaccine in healthy children and adolescents 4 to 17 years of age.

ELIGIBILITY:
Inclusion Criteria:

- Healthy subjects 4-17 years of age

Exclusion Criteria:

* Subjects who are not healthy,
* Subjects who are pregnant or breast feeding,
* Subjects with a history of severe allergic reaction or allergic to any of the vaccine components.

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2055 (Actual)
Dates: Start 2013-05; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Vaccines and Diagnostics, Study Chair — Novartis Vaccines
Locations (34):
- United States (18):
  - 320, Novartis Investigational Site, Mobile, Alabama
  - 312, Novartis Investigational Site, Ponte Vedra, Florida
  - 313, Novartis Investigational Site, Augusta, Kansas
  - 305, Novartis Investigational Site, Newton, Kansas
  - 302, Novartis Investigational Site, Wichita, Kansas
  - 301, Novartis Investigational Site, Wichita, Kansas
  - 311, Novartis Investigational Site, Fremont, Nebraska
  - 308, Novartis Investigational Site, Winston-Salem, North Carolina
  - 317, Novartis Investigational Site, Cleveland, Ohio
  - 309, Novartis Investigational Site, Tulsa, Oklahoma
  - 314, Novartis Investigational Site, Warwick, Rhode Island
  - 319, Novartis Investigational Site, Mt. Pleasant, South Carolina
  - 310, Novartis Investigational Site, Bristol, Tennessee
  - 318, Novartis Investigational Site, Nashville, Tennessee
  - 304, Novartis Investigational Site, Salt Lake City, Utah
  - 306, Novartis Investigational Site, Salt Lake City, Utah
  - 315, Novartis Investigational Site, Salt Lake City, Utah
  - 303, Novartis Investigational Site, South Jordan, Utah
- Australia (6):
  - 100, Novartis Investigational Site, Westmead, New South Wales
  - 108, Novartis Investigational Site, Auchenflower, Queensland
  - 107, Novartis Investigational Site, Sherwood, Queensland
  - 104, Novartis Investigational Site, North Adelaide, South Australia
  - 103, Novartis Investigational Site, Carlton, Victoria
  - 105, Novartis Investigational Site, Subiaco, Western Australia
- New Zealand (2):
  - 151, Novartis Investigational Site, Takapuna, Auckland
  - 150, Novartis Investigational Site, Beckenham, Christchurch
- Philippines (5):
  - 250, Novartis Investigational Site, City of Muntinlupa, Alabang
  - 251, Novartis Investigational Site, City of Muntinlupa, Alabang
  - 254, Novartis Investigational Site, City of Muntinlupa, Alabang
  - 253, Novartis Investigational Site, Manila, Ermita
  - 252, Novartis Investigation Site, Manila, Sampaloc
- Thailand (3):
  - 201, Novartis Investigational Site, Khon Kaen, Muang
  - 200, Novartis Investigational Site, Bangkok, Rajathevi
  - 202, Novartis Investigational Site, Bangkoknoi, Siriraj

REFERENCES:
- [Derived] Nolan T, Chotpitayasunondh T, Capeding MR, Carson S, Senders SD, Jaehnig P, de Rooij R, Chandra R. Safety and tolerability of a cell culture derived trivalent subunit inactivated influenza vaccine administered to healthy children and adolescents: A Phase III, randomized, multicenter, observer-blind study. Vaccine. 2016 Jan 4;34(2):230-236. doi: 10.1016/j.vaccine.2015.11.040. Epub 2015 Nov 29. PMID 26643931

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled at a total of 34 centers in 5 countries: 18 sites in the US, 6 sites in Australia, 2 sites in New Zealand, 5 sites in the Philippines and 3 sites in Thailand.
Period: Overall Study
Arm/Group | TIVc | TIVf
Started | 1372 | 683
Completed | 1359 | 673
Not Completed | 13 | 10
Not completed — ADMINISTRATIVE REASON | 0 | 1
Not completed — Lost to Follow-up | 9 | 6
Not completed — Unclassified | 3 | 3
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- TOTAL: Total of all reporting groups
Arm/Group | TIVc | TIVf | TOTAL
Number analyzed (Participants) | 1372 | 683 | 2055
Age, Continuous [Mean (Standard Deviation); unit: year] | 9.1 (3.8) | 9.3 (3.9) | 9.1 (3.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 703 | 349 | 1052
  Male | 669 | 334 | 1003

OUTCOME MEASURES:

1. Primary Outcome: Number Of Subjects Reporting Solicited Local and Systemic Adverse Events and Other Indicators Of Reactogenicity After Any Vaccination.
Description: Safety was assessed as the number of subjects who reported solicited local and systemic adverse events and other indicators of reactogenicity following two doses of either mammalian cell culture-derived or egg-derived trivalent influenza vaccination in subjects aged ≥4 To ≤17 Years.
Time Frame: Day 1 to Day 7 after any vaccination
Population: Analysis was done on the solicited safety dataset, i.e. the subjects in the exposed population who provided postvaccination solicited safety data.
Measure: Number; unit: Subjects
Groups:
- TIVc (≥4 to ≤8 Years): Subjects ≥4 to ≤8 years of age received one or two doses of mammalian cell-culture-derived trivalent influenza vaccine based on their previous vaccination status.
- TIVf (≥4 to ≤8 Years): Subjects ≥4 to ≤8 years of age received one or two doses of egg-derived trivalent influenza vaccine based on their previous vaccination status.
- TIVc (≥9 to ≤17 Years): Subjects ≥9 to ≤17 years of age received one or two doses of mammalian cell-culture-derived trivalent influenza vaccine based on their previous vaccination status.
- TIVf (≥9 to ≤17 Years): Subjects ≥9 to ≤17 years of age received one or two doses of egg-derived trivalent influenza vaccine based on their previous vaccination status.
Arm/Group | TIVc (≥4 to ≤8 Years) | TIVf (≥4 to ≤8 Years) | TIVc (≥9 to ≤17 Years) | TIVf (≥9 to ≤17 Years)
Number analyzed (Participants) | 688 | 341 | 682 | 341
Subjects
  Any Local | 422 | 202 | 370 | 160
  Injection site Induration (AE) | 109 | 43 | 46 | 33
  Injection site Swelling (AE) | 87 | 37 | 36 | 26
  Injection site Erythema (AE) | 148 | 57 | 72 | 37
  Injection site Ecchymosis (AE) | 68 | 30 | 27 | 11
  Injection site Pain (AE) | 384 | 186 | 356 | 142
  Any Systemic | 252 | 110 | 267 | 113
  Chills (AE) | 47 | 17 | 39 | 7
  Nausea (AE) | 57 | 26 | 45 | 16
  Myalgia (AE) | 113 | 41 | 126 | 44
  Arthralgia (AE) | 39 | 16 | 54 | 14
  Headache (AE) | 105 | 42 | 128 | 57
  Fatigue (AE) | 92 | 34 | 109 | 56
  Loss of appetite (AE) | 68 | 25 | 50 | 12
  Malaise (AE) | 112 | 43 | 99 | 46
  Sweating (AE) | 39 | 20 | 52 | 23
  Body Temperature (≥38°C) (AE) | 48 | 30 | 12 | 5
  ≥40°C (Other Indicator) | 3 | 0 | 0 | 0
  Prevention of pain and/or fever (Other Indicator) | 61 | 29 | 24 | 10
  Treatment of pain and/or fever (Other Indicator) | 90 | 40 | 39 | 18

2. Primary Outcome: Number Of Subjects Reporting Unsolicited Adverse Events After Any Vaccination.
Description: Safety was assessed as the number of subjects who reported unsolicited adverse events following vaccination with either mammalian cell culture-derived or egg-derived trivalent influenza vaccination in subjects aged ≥4 To ≤17 Years.
Time Frame: Day 1 to Day49 for subjects aged ≥4 To ≤8 years not previously vaccinated. Day 1 to Day 38 for subjects aged ≥4 To ≤8 years previously vaccinated and all subjects aged ≥9 To ≤17 years.
Population: Analysis was done on the unsolicited safety dataset, i.e. the subjects in the exposed population who provided postvaccination unsolicited safety data.
Measure: Number; unit: Subjects
Arm/Group | TIVc (≥4 to ≤8 Years) | TIVf (≥4 to ≤8 Years) | TIVc (≥9 to ≤17 Years) | TIVf (≥9 to ≤17 Years)
Number analyzed (Participants) | 688 | 340 | 681 | 341
Subjects
  Any AE | 277 | 139 | 158 | 88
  At least possibly related AE | 50 | 26 | 32 | 22

3. Primary Outcome: Number Of Subjects Reporting Unsolicited Serious Adverse Events After Any Vaccination.
Description: Safety was assessed as the number of subjects who reported serious adverse events (SAEs), medically attended AEs and new onset of chronic diseases (NOCD) in subjects aged ≥4 To ≤17 Years.
Time Frame: Day 1 to Day 183 for previously vaccinated subjects and Day 213 for not-previously vaccinated subjects
Population: as for outcome 2
Measure: Number; unit: Subjects
Arm/Group | TIVc (≥4 to ≤8 Years) | TIVf (≥4 to ≤8 Years) | TIVc (≥9 to ≤17 Years) | TIVf (≥9 to ≤17 Years)
Number analyzed (Participants) | 688 | 340 | 681 | 341
Subjects
  SAE | 17 | 7 | 7 | 9
  At least possibly related SAE | 0 | 0 | 0 | 0
  AE leading to withdrawal | 0 | 0 | 0 | 0
  Medically attended AE | 284 | 139 | 172 | 105
  NOCD | 5 | 4 | 3 | 1
  Death | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 6 months for subjects aged ≥4 to ≤8 years previously vaccinated and all subjects aged ≥9 to ≤17 Years 7 months for subjects aged ≥4 to ≤8 years not previously vaccinated.
Description: For subjects aged ≥4 to ≤8 years not previously vaccinated AEs collected from day 1 to 7 and day 29 to 35. SAEs, medically attended AEs and NOCD till day 213 For subjects aged ≥4 to ≤8 years previously vaccinated and subjects aged ≥9 to ≤17 Years AEs were collected from day 1 to 7. SAEs, medically attended AEs and NOCD were collected till day 183
Groups:
- TIVc(4-8Years ): Subjects ≥4 to ≤8 years of age received one or two doses of mammalian cell-culture-derived trivalent influenza vaccine based on their previous vaccination status.
- TIVf(4-8Years ): Subjects ≥4 to ≤8 years of age received one or two doses of egg-derived trivalent influenza vaccine based on their previous vaccination status.
- TIVc(9-17Years ): Subjects ≥9 to ≤17 years of age received one or two doses of mammalian cell-culture-derived trivalent influenza vaccine based on their previous vaccination status.
- TIVf(9-17Years ): Subjects ≥9 to ≤17 years of age received one or two doses of egg-derived trivalent influenza vaccine based on their previous vaccination status.
Arm/Group | TIVc(4-8Years ) | TIVf(4-8Years ) | TIVc(9-17Years ) | TIVf(9-17Years )
Serious Adverse Events (participants affected / at risk) | 17/688 | 7/341 | 7/682 | 9/341
Other Adverse Events (participants affected / at risk) | 545/688 | 267/341 | 489/682 | 220/341
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TIVc(4-8Years ) (N=688) | TIVf(4-8Years ) (N=341) | TIVc(9-17Years ) (N=682) | TIVf(9-17Years ) (N=341)
LYMPHADENITIS (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
CHOLECYSTITIS (Hepatobiliary disorders) | 0 | 0 | 1 | 0
ACUTE SINUSITIS (Infections and infestations) | 2 | 0 | 0 | 0
APPENDICITIS PERFORATED (Infections and infestations) | 1 | 0 | 0 | 0
BRONCHITIS (Infections and infestations) | 1 | 0 | 0 | 0
CELLULITIS (Infections and infestations) | 1 | 1 | 0 | 0
DENGUE FEVER (Infections and infestations) | 2 | 0 | 1 | 3
GASTROENTERITIS (Infections and infestations) | 2 | 0 | 0 | 1
NASOPHARYNGITIS (Infections and infestations) | 0 | 1 | 0 | 0
PHARYNGITIS (Infections and infestations) | 1 | 0 | 0 | 0
PHARYNGOTONSILLITIS (Infections and infestations) | 0 | 1 | 0 | 0
PNEUMONIA (Infections and infestations) | 0 | 0 | 1 | 0
RESPIRATORY SYNCYTIAL VIRUS INFECTION (Infections and infestations) | 1 | 0 | 0 | 0
SINUSITIS BACTERIAL (Infections and infestations) | 1 | 0 | 0 | 0
URINARY TRACT INFECTION (Infections and infestations) | 1 | 0 | 0 | 0
WOUND INFECTION (Infections and infestations) | 1 | 0 | 0 | 0
ANIMAL BITE (Injury, poisoning and procedural complications) | 3 | 3 | 0 | 0
ANIMAL SCRATCH (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0
HEAD INJURY (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
INJURY (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
LIGAMENT RUPTURE (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
MULTIPLE INJURIES (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
RADIUS FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
CEREBELLAR ATAXIA (Nervous system disorders) | 1 | 0 | 0 | 0
VISUAL FIELD DEFECT (Nervous system disorders) | 0 | 0 | 0 | 1
ABORTION SPONTANEOUS (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 1
ADNEXAL TORSION (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | TIVc(4-8Years ) (N=688) | TIVf(4-8Years ) (N=341) | TIVc(9-17Years ) (N=682) | TIVf(9-17Years ) (N=341)
NAUSEA (Gastrointestinal disorders) | 61 | 27 | 45 | 17
CHILLS (General disorders) | 48 | 18 | 39 | 8
FATIGUE (General disorders) | 95 | 36 | 109 | 56
INJECTION SITE ERYTHEMA (General disorders) | 164 | 68 | 85 | 43
INJECTION SITE HAEMORRHAGE (General disorders) | 69 | 30 | 27 | 11
INJECTION SITE INDURATION (General disorders) | 114 | 45 | 48 | 33
INJECTION SITE PAIN (General disorders) | 433 | 211 | 385 | 159
INJECTION SITE SWELLING (General disorders) | 95 | 43 | 41 | 29
MALAISE (General disorders) | 112 | 43 | 99 | 46
PYREXIA (General disorders) | 63 | 42 | 17 | 9
NASOPHARYNGITIS (Infections and infestations) | 36 | 17 | 21 | 15
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 133 | 60 | 58 | 26
VIRAL INFECTION (Infections and infestations) | 35 | 14 | 14 | 8
DECREASED APPETITE (Metabolism and nutrition disorders) | 68 | 25 | 51 | 12
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 41 | 16 | 57 | 15
MYALGIA (Musculoskeletal and connective tissue disorders) | 115 | 41 | 130 | 45
HEADACHE (Nervous system disorders) | 108 | 44 | 137 | 62
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 39 | 20 | 52 | 23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days